CLINICAL TRIAL: NCT03404739
Title: Single- Versus Multiple-dose Antimicrobial Prophylaxis for The Prevention of Infectious Complications Associated With Peroral Endoscopic Myotomy(POEM) for Achalasia: A Triple-Blind, Randomized Controlled, Non-Inferiority Trial
Brief Title: Single- Versus Multiple-dose Antimicrobial Prophylaxis for The Prevention of Infectious Complications Associated With Peroral Endoscopic Myotomy(POEM) for Achalasia
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: ABX for POEM
Record Dates: First submitted 2018-01-08; First posted 2018-01-19 (Actual); Last update posted 2018-11-07 (Actual); Status verified 2018-01

CONDITIONS: Esophageal Achalasia
Keywords: Antibiotic prophylaxis; Infectious complications; Peroral endoscopic myotomy
MeSH Terms: conditions — Esophageal Achalasia | interventions — Saline Solution; Ceftazidime

STUDY DESIGN:
Intervention Model Description: single- versus multiple-dose antimicrobial prophylaxis
Who Masked: Participant, Care Provider, Investigator
Masking Description: Sequentially numbered, opaque sealed envelopes(SNOSE) will be the method to conceal allocation from the study team.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Single-dose group (Experimental): Ceftazidime 2g at the start of POEM
  Interventions: Drug: Saline Solution
- Multiple-dose group (Active Comparator): Ceftazidime 2g at the start of POEM plus additional 2 doses given every 12 hours after the procedure
  Interventions: Drug: Ceftazidime

INTERVENTIONS:
Drug: Saline Solution — These patients will be given only one dose of ceftazidime at the start of POEM plus 2 doses of saline solution every 12 hours after the procedure.
  Arms: Single-dose group
Drug: Ceftazidime — These patients will be given ceftazidime 2g at the start of POEM plus additional 2 doses given every 12 hours after the procedure.
  Arms: Multiple-dose group

SUMMARY:
Peroral endoscopic myotomy is a novel, promising endoscopic technique for achalasia considering its minimal invasive characteristics and comparable efficacy to Heller myotomy. Numerous studies have focused on the efficacy, safety as well as technical aspects of POEM. However, few efforts have been made to the issue of antimicrobial prophylaxis in POEM. Postoperative prophylactic antibiotics are universally initiated on call to the operating room or at the start of POEM and consist of second-generation cephalosporins. The mean duration of antibiotic regimen after POEM was 3 days ranging from 1 day to 7 days.

Numerous studies have shown that a single dose of antibiotic prophylaxis in a variety of surgical procedures. Other studies have shown that prolonged administration of antibiotics for longer than 24 hours add no benefit in many surgeries. Prolonged use of antibiotics not only increases the costs and exposure to drug toxicity directly but also may be associated with an increased risk of acquired antibiotic resistance as well as infection with Clostridium difficile.

Thus, investigators intend to perform a prospective randomized study to confirm the validity of single-dose antimicrobial prophylaxis for the prevention of infectious complications following peroral endoscopic myotomy.

DETAILED DESCRIPTION:
This prospective randomized trial is performed to confirm the noninferiority of single-dose versus multiple-dose antimicrobial prophylaxis in terms of the incidence of infectious complications associated with peroral endoscopic myotomy. Six hundred sixty-six patients undergoing POEM for achalasia will be randomized to receive only single-dose ceftazidime (2g) or an additional 2 doses every 12 hours postoperatively (multi-dose group). POEM associated infectious complications will be assessed and recorded as regional infections, remote infections and systemic infections. Infection rate, adverse events related to antibiotics and POEM, Clavien-Dindo classification of surgical complications, length of hospital stay and efficacy of POEM will be compared. Body fluid bacterial culture will be conducted in patients suspected of infectious complications.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed of esophageal achalasia
* Patients or legal surrogates willing and competent to give informed consent and to comply with follow up visits and tests

Exclusion Criteria:

* Patients with ASA score ≥3
* Patients with indications for antibiotic prophylaxis(infective endocarditis or other conditions) as determined by the American Society for Gastrointestinal Endoscopy
* Patients who have received antibiotics in the past seven days
* Patients who have possible signs of infection during preparation for POEM
* Pregnant
* Immunodeficient patients such as severe neutropenia(<0.5x1068/l) and/or advanced hematological malignancy
* Under steroid therapy
* Patients who develop intraoperative severe adverse events including severe choking and aspiration during endotracheal intubation requiring antibiotic treatment as well as severe pneumothorax, perforation, bleeding and mucosal injury cannot be closed by clips.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 666 (Estimated)
Dates: Start 2017-10-01 (Actual); Primary Completion 2018-12 (Estimated); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
Infectious complications associated with POEM | From operation day to 4 weeks after the procedure
  Including regional, remote and systemic infections.

SECONDARY OUTCOMES:
Pathogens for causing infection | From operation day to 4 weeks after the procedure
  Body fluid will be collected and cultured in patients suspected of infectious complications
Adverse effects of antibiotics | From operation day to 4 weeks after the procedure
  Any adverse events related to ceftazidime will be recorded.
Clavien-Dindo classification of surgical complications | From operation day to 4 weeks after the procedure
  Clavien-Dindo classification of surgical complications is recorded if adverse events happen related to POEM
Length of hospital stay | From admission to discharge
  Length of hospital stay will be extracted.
Efficacy of POEM | admission to 4 weeks after POEM
  Eckardt score will be compared before and after POEM.Clinical scoring system for achalasia (Eckardt score) Score Symptom Weight loss (kg)(0-3), Dysphagia(0-3), Retrosternal pain(0-3), Regurgitation(0-3)

CONTACTS AND LOCATIONS:
Overall Officials: Ping-Hong Zhou, MD, PhD, Study Chair — Zhongshan Hospital, Fudan University, Shanghai, China
Locations (1):
- Zhongshan Hospital, Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Stavropoulos SN, Modayil RJ, Friedel D, Savides T. The International Per Oral Endoscopic Myotomy Survey (IPOEMS): a snapshot of the global POEM experience. Surg Endosc. 2013 Sep;27(9):3322-38. doi: 10.1007/s00464-013-2913-8. Epub 2013 Apr 3. PMID 23549760
- [Background] Inoue H, Minami H, Kobayashi Y, Sato Y, Kaga M, Suzuki M, Satodate H, Odaka N, Itoh H, Kudo S. Peroral endoscopic myotomy (POEM) for esophageal achalasia. Endoscopy. 2010 Apr;42(4):265-71. doi: 10.1055/s-0029-1244080. Epub 2010 Mar 30. PMID 20354937
- [Background] Imamura H, Kurokawa Y, Tsujinaka T, Inoue K, Kimura Y, Iijima S, Shimokawa T, Furukawa H. Intraoperative versus extended antimicrobial prophylaxis after gastric cancer surgery: a phase 3, open-label, randomised controlled, non-inferiority trial. Lancet Infect Dis. 2012 May;12(5):381-7. doi: 10.1016/S1473-3099(11)70370-X. Epub 2012 Jan 31. PMID 22297080
- [Background] ASGE Standards of Practice Committee; Khashab MA, Chithadi KV, Acosta RD, Bruining DH, Chandrasekhara V, Eloubeidi MA, Fanelli RD, Faulx AL, Fonkalsrud L, Lightdale JR, Muthusamy VR, Pasha SF, Saltzman JR, Shaukat A, Wang A, Cash BD. Antibiotic prophylaxis for GI endoscopy. Gastrointest Endosc. 2015 Jan;81(1):81-9. doi: 10.1016/j.gie.2014.08.008. Epub 2014 Nov 11. No abstract available. PMID 25442089
- [Background] Mohri Y, Tonouchi H, Kobayashi M, Nakai K, Kusunoki M; Mie Surgical Infection Research Group. Randomized clinical trial of single- versus multiple-dose antimicrobial prophylaxis in gastric cancer surgery. Br J Surg. 2007 Jun;94(6):683-8. doi: 10.1002/bjs.5837. PMID 17514671
- [Background] Zhang XC, Li QL, Xu MD, Chen SY, Zhong YS, Zhang YQ, Chen WF, Ma LL, Qin WZ, Hu JW, Cai MY, Yao LQ, Zhou PH. Major perioperative adverse events of peroral endoscopic myotomy: a systematic 5-year analysis. Endoscopy. 2016 Nov;48(11):967-978. doi: 10.1055/s-0042-110397. Epub 2016 Jul 22. PMID 27448052